CLINICAL TRIAL: NCT04488549
Title: DElayed COloRectal Cancer Care During Coronavirus Disease (COVID-19) Pandemic (DECOR-19)
Acronym: DECOR-19
Status: Completed | Type: Observational
Sponsor: Treviso Regional Hospital (Network)
Collaborators: Gaetano Gallo (Unknown); Gian Luca Di Tanna (Unknown)
Responsible Party: Sponsor
Other Study IDs: Treviso
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Colo-rectal Cancer; Colon Cancer; Rectal Cancer; Oncology; Surgery
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — International E-survey

SUMMARY:
To understand and analyse the global impact of COVID-19 on outpatient services, inpatient care, elective surgery, and perioperative colorectal cancer care, a DElayed COloRectal cancer surgery (DECOR-19) survey was conducted in collaboration with numerous international colorectal societies with the objective of obtaining several learning points from the impact of the COVID-19 outbreak on our colorectal cancer patients which will assist us in the ongoing management of our colorectal cancer patients and to provide us safe oncological pathways for future outbreaks.

ELIGIBILITY:
Inclusion Criteria:

* Members of renowned scientific societies with an interest in coloproctology

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The survey link was sent to scientific societies of interest to coloproctologists and disseminated to their members. Participation was entirely voluntary with no compensation offered. Informed consent was obtained from all those agreeing to complete a survey. This study was exempt from review board approval at authors' institutions.
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Predictive power of respondents' and hospitals' demographics on delaying colorectal cancer care across 6 geographical regions | 20 days
  Respondents' and hospitals' demographics include: gender, country of origin, type of hospital (i.e. academic or not), type of unit (general surgery vs. colorectal), no. hospital beds, no. yearly surgeries for colon and rectal cancer, hospital preparedness to the emergency (i.e. fully or partially dedicated or not involved in COVID-19 care), readily availability of external facilities for colorectal cancer surgery, cancer care coordinator, personal protective equipment, status of elective surgery, no. elective colorectal cancer patients needing urgent surgery, any change in the original management plan, no. colorectal cancer patients refusing surgery or being COVID-19 + on surgery or becoming COVID-19 + post-operatively, no. staff members quarantined or relocated in COVID-19 units, MDT meeting suspension, any delay in endoscopy, radiology, oncology, surgery, histopathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Treviso Regional Hospital, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Undecided